CLINICAL TRIAL: NCT04242654
Title: A Randomized-Controlled Trial of Handheld Doppler Ultrasound Compared With Auscultation by Stethoscope to Assess Heart Rate During the Resuscitation of High-risk Neonates
Brief Title: Doppler Ultrasound Compared With Stethoscope to Assess Heart Rate (HR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAS5205
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Neonatal Resuscitation
Keywords: Doppler ultrasound; heart rate; neonatal resuscitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doppler ultrasound (Experimental): Placement of Doppler US on chest to obtain newborn's heart rate.
  Interventions: Procedure: Handheld fetal doppler ultrasound
- Stethoscope (No Intervention): Placement of stethoscope on chest to obtain newborn's heart rate.

INTERVENTIONS:
Procedure: Handheld fetal doppler ultrasound — Handheld fetal doppler ultrasound will be used to assess heart rate in high-risk neonates.
  Arms: Doppler ultrasound

SUMMARY:
This is a prospective randomized controlled trial comparing heart rate measurement by Doppler ultrasound or auscultation with a stethoscope in newborn infants who require stabilization or resuscitation immediately after birth. Enrolled subjects will be randomly assigned to have their heart rate (HR) obtained by stethoscope (ST) or by Doppler ultrasound (DO). Neonates will be resuscitated in accordance with the Neonatal Resuscitation Program (NRP) guidelines.

DETAILED DESCRIPTION:
Obtaining a baby's heart rate (HR) is an important part of neonatal resuscitation in the delivery room and helps the medical team decide how to treat the baby. When babies do not breathe well on their own, the medical team places electrocardiogram (ECG) leads on the baby's chest to obtain an accurate HR rapidly that can be seen by the entire team. Before the ECG leads are placed on the baby's chest, the Neonatal Resuscitation Program (NRP) guidelines suggest that medical team members listen to the baby's HR using a stethoscope for 6 seconds. However, it can take longer than 6 seconds for medical team members to obtain a HR which can delay a baby's care. The purpose of this study is to determine if Doppler ultrasound is a useful, alternative tool, aside from a stethoscope, that can be used to quickly obtain a baby's HR, particularly in high-risk babies. The primary objective will be the time that it takes to obtain a baby's HR by Doppler ultrasound as compared to listening to a baby's HR with a stethoscope. With this study, the investigators will be able to understand if Doppler ultrasound is a useful tool in the resuscitation of babies who are high risk.

ELIGIBILITY:
Inclusion Criteria:

* All neonates admitted to the transitional nursery for resuscitation after delivery

Exclusion Criteria:

* Neonates with congenital heart disease, congenital diaphragmatic hernia
* Neonates whose mothers present and will have imminent delivery

Ages: 0 Hours to 1 Hour | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Time to obtain HR (in seconds) | Up to approximately 1 minute
  The primary outcome will be the time to obtain heart rate (HR), which will be defined as the time from when the neonate is placed on the radiant warmer to the time the HR is indicated to the entire resuscitation team.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Leone A. Leone, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No